CLINICAL TRIAL: NCT06463756
Title: CT-based Radiomics, Two-dimensional and Three-dimensional Deep Learning Models to Predict Thyroid Cartilage Invasion in Laryngeal Carcinoma: a Multicenter Study
Brief Title: AI Models to Predict Thyroid Cartilage Invasion in Laryngeal Carcinoma
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Collaborators: Nankai University (Other)
Responsible Party: Principal Investigator, xinwei Chen, Radiology Department, First Affiliated Hospital of Chongqing Medical University
Other Study IDs: 2024-Chenx
Record Dates: First submitted 2024-06-12; First posted 2024-06-18 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Laryngeal Carcinoma; Thyroid Cartilage
Keywords: radiomics; deep learning
MeSH Terms: conditions — Laryngeal Neoplasms | interventions — Deep Learning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- training cohort: No interventions
  Interventions: Other: AI
- internal validation cohort: No interventions
  Interventions: Other: AI
- external validation cohort: No interventions
  Interventions: Other: AI

INTERVENTIONS:
Other: AI — Radiomics extracts quantitative information from medical images to generate high-dimensional feature vectors for analysis. It aims to provide insights into disease processes and improve diagnosis.
  Deep learning utilizes neural networks with multiple layers to learn complex patterns from data. In medical imaging, it enables accurate and efficient analysis for disease detection and diagnosis.
  Other Names: radiomics; deep learning

SUMMARY:
This retrospective study was to develop and verify CT-based AI model to preoperatively predict the thyroid cartilage invasion of laryngeal cancer patients, so as to provide more accurate diagnosis and treatment basis for clinicians. In addition, the researchers investigated the prediction of survival outcomes of patients by the above optimal models.

DETAILED DESCRIPTION:
Laryngeal squamous cell carcinoma (LSCC), as one of the most common head and neck tumors, is the eighth leading cause of cancer-associated death worldwide. The treatment decisions has a profound impact on both tumor control and functional prognosis of LSCC patients. And these decisions are primarily based on tumor staging, with the invasion of the thyroid cartilage serving as a crucial determinant. Consequently, the presence of thyroid cartilage invasion indicates an advanced stage (T3 or T4) diagnosis for the LSCC patients. For patients without thyroid cartilage invasion, partial laryngectomy may be considered to preserve laryngeal function. However, for patients with advanced laryngeal carcinoma and thyroid cartilage invasion extending beyond the larynx, total laryngectomy is often necessary to completely remove the tumor and extend survival time. Therefore, accurate assessment of thyroid cartilage invasion is vital for treatment decision-making and prognosis evaluation for LSCC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Availability of complete clinical data
2. Surgery-proven or biopsy-proven diagnosis of laryngeal squamous cell carcinoma
3. CT examination performed within 2 weeks before surgery

Exclusion Criteria:

1. Patients who received preoperative chemotherapy or radiation therapy
2. CT images with significant artifacts
3. Patients with tumor recurrence

Ages: 18 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators collected patients with laryngeal carcinoma from two centers.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-08-13 (Actual); Primary Completion 2024-09-13 (Estimated); Study Completion 2024-10-13 (Estimated)

PRIMARY OUTCOMES:
Area under the curve, AUC | Through study completion, an average of 6 months
  Area under the curve(AUC) is a metric widely used in machine learning and medical research to evaluate the performance of models in binary classification problems. It reflects the ability of a model to identify true positives (True Positives) while avoiding falsely classifying negative examples as positive (False Positives).

SECONDARY OUTCOMES:
Disease-Free-Survival, DFS | The date of surgery and the occurrence of events such as disease progression, the date of the last follow-up, or death from any cause, and the follow-up time was at least 3 years
  Disease-Free Survival (DFS) refers to the time from the start of randomization (usually the starting point of a clinical trial) to the recurrence of the disease or death of the patient due to disease progression. DFS is an important clinical and statistical indicator used to evaluate the long-term effects of cancer treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, China

IPD SHARING:
Plan to Share IPD: No
The clinical data are manually collected from the clinical case system; the CT image data are exported from the PACS system and anonymously stored on a separate data disk; and the image materials are collected and anonymously stored on a separate data disk.